CLINICAL TRIAL: NCT01148979
Title: Double-Blind, Placebo-Controlled, Randomized Trial of Adjunctive Lisdexamfetamine Dimesylate in Residual Symptoms of Major Depressive Disorder Partially Responsive to Selective Serotonin or Norepinephrine Reuptake Inhibitor Monotherapy
Brief Title: Lisdexamfetamine Dimesylate in Residual Symptoms and Cognitive Impairment in Major Depressive Disorder.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: Shire (Industry)
Responsible Party: Principal Investigator, J. Alexander Bodkin, Director, Clinical Psychopharmacology Research Program, Mclean Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2010-P-000871
Record Dates: First submitted 2010-06-21; First posted 2010-06-23 (Estimated); Results first posted 2017-05-23 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-04

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Cognitive Impairment; Partial Response; Residual Symptoms
MeSH Terms: conditions — Depressive Disorder, Major; Cognitive Dysfunction | interventions — Lisdexamfetamine Dimesylate; Sugars

STUDY DESIGN:
Intervention Model Description: This is a double-blind, placebo-controlled, crossover study in which each subject will act as their own control after being randomly assigned to placebo or Lisdexamfetamine Dimesylate (Vyvanse) for the first 4 weeks of study treatment, then receiving the other for the second 4 weeks of treatment. The two 4-week treatment periods are separated by a washout of 2 weeks.
Who Masked: Participant, Investigator
Masking Description: Both the study participant and the study investigators making evaluations are blinded to which treatment arm the participants are assigned to (i.e., whether they are receiving placebo or Vyvanse at any given point). Placebo and active medication capsules look identical.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adjunct Lisdexamfetamine (Vyvanse) (Experimental): Participants receive Lisdexamfetamine Dimesylate 20-50 mg capsule each morning for 4 weeks. After a washout period of 2 weeks, they receive Placebo capsule (matching Lisdexamfetamine Dimesylate (Vyvanse) capsule) each morning for 4 weeks.
  Interventions: Drug: Lisdexamfetamine Dimesylate (Vyvanse)
- Adjunct Placebo (Placebo Comparator): Participants receive Placebo capsule (matching Lisdexamfetamine Dimesylate (Vyvanse) 20-50 mg capsule) each morning for 4 weeks. After a washout period of 2 weeks, they receive Lisdexamfetamine Dimesylate capsule each morning for 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lisdexamfetamine Dimesylate (Vyvanse) — Lisdexamfetamine Dimesylate (Vyvanse) capsules dose ranging from 20mg to 50 mg.
  Other Names: Vyvanse
  Arms: Adjunct Lisdexamfetamine (Vyvanse)
Drug: Placebo — Lisdexamfetamine Dimesylate (Vyvanse)-matched placebo capsules.
  Other Names: Sugar pill
  Arms: Adjunct Placebo

SUMMARY:
This study aims to test the effect of a newly-approved stimulant medication, lisdexamfetamine dimesylate (Vyvanse), on specific residual symptoms of depression found in some patients who are undergoing treatment with, but have only partially responded to, a selective-serotonin reuptake inhibitor (SSRI) or selective-norepinephrine reuptake inhibitor (SNRI) antidepressant. Specifically, the investigators hypothesize that symptoms potentially related to deficient dopaminergic activity, such as lassitude, apathy, reduced positive affect and impaired executive function, in particular, will improve. This protocol is designed to test the hypothesis that this cluster of co-occurring residual symptoms sometimes found in treated depression will respond as a group to adjunctive psychostimulant therapy. The investigators propose to demonstrate this cluster of residual depressive symptoms and to measure the effect of stimulant therapy on it. The investigators hope to better understand the specific symptoms in this clinical population that are likely to improve with stimulant therapy.

DETAILED DESCRIPTION:
This protocol is designed to test the hypothesis that a cluster of co-occurring residual symptoms sometimes found in treated depression will respond as a group to psychostimulant therapy. This cluster includes apathy, reduced drive, fatigue, impaired executive function and other cognitive measures, and low positive affect. We propose to measure this cluster of symptoms in a population of residually depressed subjects demonstrating them, and then to measure the effect of stimulant therapy on this cluster, and each constituent symptom, as well as to measure its effect on subjects' overall functional impairment, and to document treatment emergent adverse effects. The goal is to gather data about the response of these residual symptoms to stimulant therapy. Since each subject will be exposed to active treatment and matched placebo, a benefit to individual participants will be to learn if their specific symptom burden is ameliorated by stimulant therapy, and what adverse effects may emerge for them. We hope to develop an understanding of the specific symptoms in this clinical population that are likely to improve with stimulant therapy. We also hope to be able to characterize the side effect burden of stimulant therapy in this clinical population.

ELIGIBILITY:
Inclusion Criteria:

1. Meeting diagnostic criteria for major depression during the present episode of illness, currently with at least mild improvement by report (CGI-I ≥3) but with continuing residual symptoms.
2. A score of ≥10 on MADRS items 1,2,6,7 and 8, (the MADRS Dysphoric Apathy/Retardation factor, Parker et al., 2003) at screening and randomization. These 5 items are: Apparent sadness, Reported sadness, Concentration difficulties, Lassitude, and Inability to feel. A score of ≥3 will be required for at least 2 of these items.
3. A score of 3 or 4 on the Clinical Global Impression of Severity (CGI-S) at screening and randomization.
4. At randomization subjects must have received therapeutic dosages of approved SSRI or SNRI agents for at least 8 weeks, with the last 4 weeks at a constant dosage.
5. Females of Child-bearing Potential (FOCP) must have a negative serum beta Human Chorionic Gonadotropin (B-hCG) pregnancy test at the screening visit and a negative urine pregnancy test at the baseline visit, and agree to use one of the following methods of birth control: oral contraceptives, contraceptive implants, injectable contraceptives, IUDs, double-barrier contraception, sexual abstinence or vasectomized partner(s).

Exclusion Criteria:

1. Treatment within 4 weeks of randomization with any non-SSRI/SNRI antidepressant (trazodone is permitted up to 100 mg at night for sleep); any antipsychotic agent; any mood stabilizer; any standing benzodiazepine regimen other than at low doses for sleep (≤ 1 mg lorazepam HS or the equivalent); or a standing regimen of any other agent that may affect cognitive function (e.g., psychostimulants, including modafinil or R-modafinil).
2. Any current or past psychotic disorder, Bipolar I or II disorder, Current panic disorder, History of ADHD, Antisocial Personality Disorder or Borderline Personality Disorder, Mental retardation or any dementing disorder.
3. Covi Anxiety Scale score greater than Raskin Depression Scale score at Screening, to exclude subjects with more prominent anxiety than depression
4. MADRS Sleep (item 4), or Appetite (item 5) >3 at screening or randomization
5. Initial insomnia at screening that is not adequately controlled by sleep medication (trazodone up to 100 mg HS for sleep and/or ≤ 1 mg lorazepam HS or the equivalent).
6. Medical conditions that might be exacerbated by Vyvanse treatment, such as uncontrolled hypertension or angina; or conditions that would make study findings hard to interpret, such as hyperthyroidism
7. History of seizure (other than infantile febrile seizures), any tic disorder, or a current diagnosis and/or family history of Tourette's Disorder.
8. Known cardiac structural abnormality or any other condition that may affect cardiac performance
9. Any clinically significant ECG or laboratory abnormality at Screening
10. Current abnormal thyroid function, as defined by abnormal TSH at Screening (Treatment with a stable dose of thyroid medication for at least 3 months is permitted if TSH is normal at screening).
11. Suicide attempt within the past 2 years or a history of any homicidal behavior.
12. MADRS Suicidal thoughts (item 10) >4 at any study visit, or if a patient is considered by the investigator to be at clinical risk of suicide at any time in the course of the study.
13. resting sitting systolic blood pressure >149mmHg or diastolic blood pressure > 95mmHg. Subjects may be on monotherapy with anti-hypertensive medication.
14. documented allergy, hypersensitivity, intolerance, or non-responsivity to methylphenidate or amphetamines.
15. Subject has a history of a substance use disorder (abuse or dependence, as defined by DSM-IV-TR™), with the exception of nicotine dependence, within 6 months prior to screening.
16. Subject has glaucoma
17. Subject is taking other medications that have central nervous system (CNS) effects or affect performance, such as sedating antihistamines and decongestant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-09; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Alexander Bodkin Bodkin, MD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bodkin JA, Lasser RA, Wines JD Jr, Gardner DM, Baldessarini RJ. Combining serotonin reuptake inhibitors and bupropion in partial responders to antidepressant monotherapy. J Clin Psychiatry. 1997 Apr;58(4):137-45. doi: 10.4088/jcp.v58n0401. PMID 9164423
- [Background] Candy M, Jones L, Williams R, Tookman A, King M. Psychostimulants for depression. Cochrane Database Syst Rev. 2008 Apr 16;(2):CD006722. doi: 10.1002/14651858.CD006722.pub2. PMID 18425966
- [Background] Dunkin JJ, Leuchter AF, Cook IA, Kasl-Godley JE, Abrams M, Rosenberg-Thompson S. Executive dysfunction predicts nonresponse to fluoxetine in major depression. J Affect Disord. 2000 Oct;60(1):13-23. doi: 10.1016/s0165-0327(99)00157-3. PMID 10940443
- [Background] Edgar CJ, Pace-Schott EF, Wesnes KA. Approaches to measuring the effects of wake-promoting drugs: a focus on cognitive function. Hum Psychopharmacol. 2009 Jul;24(5):371-89. doi: 10.1002/hup.1034. PMID 19565524
- [Background] Fava M, Graves LM, Benazzi F, Scalia MJ, Iosifescu DV, Alpert JE, Papakostas GI. A cross-sectional study of the prevalence of cognitive and physical symptoms during long-term antidepressant treatment. J Clin Psychiatry. 2006 Nov;67(11):1754-9. doi: 10.4088/jcp.v67n1113. PMID 17196056
- [Background] Fava M, Thase ME, DeBattista C. A multicenter, placebo-controlled study of modafinil augmentation in partial responders to selective serotonin reuptake inhibitors with persistent fatigue and sleepiness. J Clin Psychiatry. 2005 Jan;66(1):85-93. doi: 10.4088/jcp.v66n0112. PMID 15669893
- [Background] Fleurence R, Williamson R, Jing Y, Kim E, Tran QV, Pikalov AS, Thase ME. A systematic review of augmentation strategies for patients with major depressive disorder. Psychopharmacol Bull. 2009;42(3):57-90. PMID 19752841
- [Background] Gorlyn M, Keilp JG, Grunebaum MF, Taylor BP, Oquendo MA, Bruder GE, Stewart JW, Zalsman G, Mann JJ. Neuropsychological characteristics as predictors of SSRI treatment response in depressed subjects. J Neural Transm (Vienna). 2008 Aug;115(8):1213-9. doi: 10.1007/s00702-008-0084-x. Epub 2008 Jul 16. PMID 18629432
- [Background] Parker RD, Flint EP, Bosworth HB, Pieper CF, Steffens DC. A three-factor analytic model of the MADRS in geriatric depression. Int J Geriatr Psychiatry. 2003 Jan;18(1):73-7. doi: 10.1002/gps.776. PMID 12497559
- [Background] Ravindran AV, Kennedy SH, O'Donovan MC, Fallu A, Camacho F, Binder CE. Osmotic-release oral system methylphenidate augmentation of antidepressant monotherapy in major depressive disorder: results of a double-blind, randomized, placebo-controlled trial. J Clin Psychiatry. 2008 Jan;69(1):87-94. doi: 10.4088/jcp.v69n0112. PMID 18312042
- [Background] Taylor BP, Bruder GE, Stewart JW, McGrath PJ, Halperin J, Ehrlichman H, Quitkin FM. Psychomotor slowing as a predictor of fluoxetine nonresponse in depressed outpatients. Am J Psychiatry. 2006 Jan;163(1):73-8. doi: 10.1176/appi.ajp.163.1.73. PMID 16390892
- [Background] Trivedi MH, Rush AJ, Wisniewski SR, Nierenberg AA, Warden D, Ritz L, Norquist G, Howland RH, Lebowitz B, McGrath PJ, Shores-Wilson K, Biggs MM, Balasubramani GK, Fava M; STAR*D Study Team. Evaluation of outcomes with citalopram for depression using measurement-based care in STAR*D: implications for clinical practice. Am J Psychiatry. 2006 Jan;163(1):28-40. doi: 10.1176/appi.ajp.163.1.28. PMID 16390886

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 35 potential subjects were screened for eligibility between September 2010 and April 2014 at McLean Hospital in Belmont, MA.
Pre-assignment Details: Of the 35 subjects screened, 29 were randomized. Of the 6 not randomized, 3 did not meet inclusion criteria, 1 withdrew consent, and 2 were lost to follow post screening. Of the 29 randomized, 28 completed both parts of the study. One subject was lost to follow after 3 weeks in the first half. Data were analyzed for the 28 completers only.
Groups:
- Placebo, Then Vyvanse: Participants first received Placebo capsule (matching Lisdexamfetamine Dimesylate(Vyvanse) 20-50 mg capsule) each morning for 4 weeks. After a washout period of 2 weeks, they then received Lisdexamfetamine Dimesylate (Vyvanse) capsule each morning for 4 weeks, starting with initial dose 30 mg/d.
  Lisdexamfetamine Dimesylate (Vyvanse): Lisdexamfetamine Dimesylate (Vyvanse) capsules dose ranging from 20mg to 50 mg.
  Placebo: Lisdexamfetamine Dimesylate (Vyvanse)-matched placebo capsules.
- Vyvanse, Then Placebo: Participants first received Lisdexamfetamine Dimesylate (Vyvanse) 20-50 mg capsule each morning for 4 weeks, staring with initial dose 30 mg/d. After a washout period of 2 weeks, they then received Placebo capsule (matching Lisdexamfetamine Dimesylate (Vyvanse) capsule) each morning for 4 weeks.
  Lisdexamfetamine Dimesylate (Vyvanse): Lisdexamfetamine Dimesylate (Vyvanse) capsules dose ranging from 20mg to 50 mg.
  Placebo: Lisdexamfetamine Dimesylate (Vyvanse)-matched placebo capsules.
Period: Overall Study
Arm/Group | Placebo, Then Vyvanse | Vyvanse, Then Placebo
Started | 13 | 16
Completed | 13 | 15
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo, Then Vyvanse: Participants first received Placebo capsule (matching Lisdexamfetamine Dimesylate(Vyvanse) 20-50 mg capsule) each morning for 4 weeks. After a washout period of 2 weeks, they then received Lisdexamfetamine Dimesylate capsule each morning for 4 weeks.
  Lisdexamfetamine Dimesylate (Vyvanse): Lisdexamfetamine Dimesylate (Vyvanse) capsules dose ranging from 20mg to 50 mg.
  Placebo: Lisdexamfetamine Dimesylate (Vyvanse)-matched placebo capsules.
- Vyvanse, Then Placebo: Participants first received Lisdexamfetamine Dimesylate 20-50 mg capsule each morning for 4 weeks. After a washout period of 2 weeks, they then received Placebo capsule (matching Lisdexamfetamine Dimesylate (Vyvanse) capsule) each morning for 4 weeks.
  Lisdexamfetamine Dimesylate (Vyvanse): Lisdexamfetamine Dimesylate (Vyvanse) capsules dose ranging from 20mg to 50 mg.
  Placebo: Lisdexamfetamine Dimesylate (Vyvanse)-matched placebo capsules.
- Total: Total of all reporting groups
Arm/Group | Placebo, Then Vyvanse | Vyvanse, Then Placebo | Total
Number analyzed (Participants) | 13 | 16 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.8 (10.6) | 48.9 (11.4) | 50.6 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 8 | 9 | 17
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 16 | 29

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Dysphoric Apathy/Retardation Sub-factor (MDAR) of Montgomery-Asberg Depression Rating Scale (MADRS) at 4 Weeks.
Description: The Montgomery-Asberg Depression Rating Scale Dysphoric Apathy Retardation subfactor (MDAR) is a 5-item subscale of the clinician-administered 10-item Montgomery-Asberg Depression Rating Scale (MADRS). MDAR score can range from 0-30 with a higher score representing a greater severity of depressive symptoms.
Time Frame: Baseline to 4 weeks of treatment
Population: All participants who completed all 4 weeks on both treatments (i.e., Placebo and Vyvanse) were included in the analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Placebo Adjunct: Participants first received Placebo capsule (matching Lisdexamfetamine Dimesylate(Vyvanse) 20-50 mg capsule) each morning for 4 weeks. After a washout period of 2 weeks, they then received Lisdexamfetamine Dimesylate (Vyvanse) capsule each morning for 4 weeks, starting with initial dose 30 mg/d.
  Lisdexamfetamine Dimesylate (Vyvanse): Lisdexamfetamine Dimesylate (Vyvanse) capsules dose ranging from 20mg to 50 mg.
  Placebo: Lisdexamfetamine Dimesylate (Vyvanse)-matched placebo capsules.
- Lisdexamfetamine Dimesylate (Vyvanse): Participants first received Lisdexamfetamine Dimesylate (Vyvanse) 20-50 mg capsule each morning for 4 weeks, staring with initial dose 30 mg/d. After a washout period of 2 weeks, they then received Placebo capsule (matching Lisdexamfetamine Dimesylate (Vyvanse) capsule) each morning for 4 weeks.
  Lisdexamfetamine Dimesylate (Vyvanse): Lisdexamfetamine Dimesylate (Vyvanse) capsules dose ranging from 20mg to 50 mg.
  Placebo: Lisdexamfetamine Dimesylate (Vyvanse)-matched placebo capsules.
Arm/Group | Placebo Adjunct | Lisdexamfetamine Dimesylate (Vyvanse)
Number analyzed (Participants) | 13 | 15
scores on a scale
  Baseline Mean MDAR score | 12.57 (3.98) | 13.46 (3.94)
  Week 4 Mean MDAR score | 9.08 (5.51) | 6.36 (5.54)
  Change from BL in mean MDAR score | -3.49 (4.66) | -7.08 (5.03)
Statistical Analysis 1: Comparison: Placebo Adjunct vs Lisdexamfetamine Dimesylate (Vyvanse); The statistical analysis represents a within-subject comparison of change under treatment with Vyvanse versus change under treatment with placebo, using paired t-tests with each subject as their own control. All tests reported are two-tailed; Test type: Other — A Paired sample t-test was used to test the null hypothesis of no difference in MDAR score change after 4 weeks of treatment with Vyvanse versus placebo; p < 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the 4 years of active subject participation.
Arm/Group | Adjunct Lisdexamfetamine (Vyvanse) | Adjunct Placebo
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 23/28 | 18/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adjunct Lisdexamfetamine (Vyvanse) (N=28) | Adjunct Placebo (N=28)
decreased appetite (General disorders) | 8 | 2
headache (General disorders) | 3 | 5
dry mouth (General disorders) | 7 | 1
insomnia (General disorders) | 10 | 3
irritability (Psychiatric disorders) | 3 | 0
anxiety (Psychiatric disorders) | 4 | 4
upper respiratory infection (Infections and infestations) | 1 | 2
fatigue (General disorders) | 1 | 2
gastrointesinal disturbance (Gastrointestinal disorders) | 1 | 4
increased activation (Psychiatric disorders) | 0 | 2
diaphoresis (General disorders) | 2 | 1 — increased sweating
decreased libido (General disorders) | 2 | 1
stomach virus (Infections and infestations) | 0 | 3
tinnitus (Nervous system disorders) | 2 | 0
muscle tension (Musculoskeletal and connective tissue disorders) | 4 | 0
tachycardia (Cardiac disorders) | 3 | 0
paresthesia (Nervous system disorders) | 2 | 0

LIMITATIONS AND CAVEATS:
The small sample size and crossover design both weaken group differences.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No